CLINICAL TRIAL: NCT05211115
Title: Randomised Clinical Trial Comparing Autogenous vs. Xenogeneic Peri-implant Soft Tissue Grafts Placed in Full vs. Split Thickness Flaps: a Clinical, Histological and Vascular Analysis
Brief Title: Autogenous vs. Xenogeneic Peri-implant Soft Tissue Grafts Placed in Full vs. Split Thickness Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-102
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2023-05

CONDITIONS: Thin Gingiva
Keywords: Soft tissue management; Dental implant; Collagen matrix; Connective tissue graft; Split thickness flap; Full thickness flap

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Split thickness flap + Volume stable collagen matrix (Experimental): A split thickness flap will be raised with a micro-blade, keeping a flap thickness >0,5mm. The healing abutment will be connected to the implant, and a 10mm wide, 6-8mm high, 6mm thick volume stable collagen matrix will be stabilised at the inner aspect of the flap.
  Interventions: Procedure: Split thickness flap; Procedure: Volume stable collagen matrix
- Full thickness flap + Volume stable collagen matrix (Active Comparator): A full thickness flap will be raised with a periosteal elevator. The healing abutment will be connected to the implant, and a 10mm wide by 6-8mm high volume stable collagen matrix will be stabilised at the inner aspect of the flap.
  Interventions: Procedure: Full thickness flap; Procedure: Volume stable collagen matrix
- Split thickness flap + Autogenous connective tissue (Active Comparator): A split thickness flap will be raised with a micro-blade, keeping a flap thickness >0,5mm. The healing abutment will be connected to the implant, and a 10mm wide, 6-8mm high, 1,5mm thick autogenous sub epithelial connective tissue graft will be stabilised at the inner aspect of the flap.
  Interventions: Procedure: Split thickness flap; Procedure: Autogenous sub epithelial connective tissue graft
- Full thickness flap + Autogenous connective tissue (Active Comparator): A full thickness flap will be raised with a periosteal elevator. The healing abutment will be connected to the implant, and a 10mm wide, 6-8mm high, 1,5mm thick autogenous sub epithelial connective tissue graft will be stabilised at the inner aspect of the flap.
  Interventions: Procedure: Full thickness flap; Procedure: Autogenous sub epithelial connective tissue graft

INTERVENTIONS:
Procedure: Split thickness flap — Palatally displaced crestal incision at the edentulous site, combined with the split thickness elevation of a buccal flap, extended to the sulcus of the adjacent mesial and distal tooth. Flap elevation performed with a micro-blade, in a buccal and apical direction, for approximately 15mm apical to the crestal incision.
  Arms: Split thickness flap + Autogenous connective tissue; Split thickness flap + Volume stable collagen matrix
Procedure: Full thickness flap — Palatally displaced crestal incision at the edentulous site, combined with the full thickness elevation of a buccal flap, extended to the sulcus of the adjacent mesial and distal tooth. Flap elevation performed with a fine periosteal elevator, in a buccal and apical direction, for approximately 15mm apical to the crestal incision.
  Arms: Full thickness flap + Autogenous connective tissue; Full thickness flap + Volume stable collagen matrix
Procedure: Autogenous sub epithelial connective tissue graft — Harvest of a sub epithelial connective tissue graft using a double incision technique, approximately 2-3 mm apical to the palatal gingival margins of the first and second premolars. Graft dimension standardised as 10mm (mesio-distally) by 6-8mm (apico-coronally) by 1,5mm (thickness). Graft stabilised at the inner aspect of the buccal flap, 1mm apical to the flap margin, using one mesial and one distal horizontal mattress sutures.
  Arms: Full thickness flap + Autogenous connective tissue; Split thickness flap + Autogenous connective tissue
Procedure: Volume stable collagen matrix — Geistlich Fibro-Gide® matrix shaped at a standardised dimension of 10mm (mesio-distally) by 6-8mm (apico-coronally) by 6mm (thickness). Matrix stabilised at the inner aspect of the buccal flap, 1mm apical to the flap margin, using one mesial and one distal horizontal mattress sutures.
  Arms: Full thickness flap + Volume stable collagen matrix; Split thickness flap + Volume stable collagen matrix

SUMMARY:
Randomized, outcome assessor and data analyst blinded, single center trial with four parallel arms and a 1:1:1:1 allocation ratio, with the aim of comparing which combination of bilaminar technique (split vs. full thickness flap) and graft type (autogenous or xenogeneic) provides better clinical, aesthetic, morphological, vascular and patients related outcomes, when augmenting the buccal peri-implant mucosa at the reopening of submerged implant fixtures

DETAILED DESCRIPTION:
This randomized four parallel arms controlled clinical trial with blinded outcome assessment and data analysis aims to establish which combination of bilaminar technique (split vs. full thickness flap) and graft type (autogenous subepithelial connective tissue graft vs. volume stable collagen matrix) provides better clinical, aesthetic, morphological, vascular and patients related outcomes, when augmenting the buccal peri-implant mucosa at the reopening of submerged implant fixtures. The primary outcome is the gain in soft tissue thickness (standardised measurement at baseline, after surgery, at 1m and 6m). Secondary outcomes include changes in tissue volume (intraoral scans at baseline, post-op, 14d, 1m, 6m), RAL and KTW (clinical measurements at baseline, 1m, 6m), tissue color integration (∆E at 1m and 6m), and PROMS (7d, 14d, 30d). Exploratory outcomes include tissue morphology (histology at 1m,2m,4m,6m), microcirculation (Doppler flowmetry at pre-op, 7d, 14d, 1m) and revascularization (IHC at 1m,2m,4m,6m). A figure of 10 subjects per group was obtained for a 0,3mm difference in tissue thickness increase (SD 0,23mm), using 80% power, alpha 0.05, and a 10% drop-out rate. Patients will be randomly allocated to four groups: test (STF+VCM), control 1 (FTF+VCM), control 2 (SFT+CTG), control 3 (FTF+CTG). Patients will be the unit of analysis and ANOVA (normality) or Kruskall-Wallis (no normality) tests will be performed setting the significance level at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Any male or female adult (≥ 18 year old) patient from the University Complutense of Madrid, being able to sign an informed consent form, presenting a submerged dental implant scheduled to undergo a second stage surgery, which is bounded mesially or distally by a remaining natural tooth, and exhibits a lack of buccal soft tissue volume, will be potentially eligible for this trial.

The case definition for a lack of buccal soft tissue volume will be the presence of a thin buccal mucosa (< 2mm) or a minor volumetric contraction of the alveolar process (flat or concave buccal mucosal profile at the edentulous area).

Exclusion Criteria:

Patients fitting to all the above inclusion criteria will be not included in the study if unable to attend to the study-related procedures (including the follow-up visits) or if one or more of the following systemic or local exclusion criteria will be found during enrolment or through the study:

Systemic primary exclusion criteria:

* Compromised general health status contraindicating the study procedures (≥ASA IV);
* Drug abuse, alcohol abuse, or smoking > 10 cigarettes a day;
* Chronic use of corticosteroids, NSAIDs, or immune-modulators (any type, any dose);
* Assumption of bisphosphonates (any type, any dose, past or present);
* Pregnant or nursing women;
* Hypersensitivity to paracetamol;

Local primary exclusion criteria

* History of previous mucogingival surgeries in the area of interest;
* Lack of adequate vestibule depth to perform a bilaminar procedure;
* Lack of osseointegration at the time of implant reopening;
* Need for additional bone grafting at the time of implant reopening;
* Intraoperative evidence of a flap thickness < 0,5mm or > 2mm.

Secondary exclusion criteria:

- Non compliant patients: poor oral hygiene at 2 consecutive visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Buccal soft tissue thickness | before surgery, after surgery, 1 month after surgery, 6 months after surgery
  Changes in the thickness of the buccal peri-implant mucosa, measured with trans-gingival probing.

SECONDARY OUTCOMES:
Volume changes | before surgery, after surgery, 14 days after surgery, 1 month after surgery, 6 months after surgery
  Changes in the size of the buccal peri-implant tissues and in their volume distribution, measured with a digital volumetric analysis.
Attachment level | baseline, after surgery, 1 month after surgery, 6 months after surgery
  Relative attachment level (implant) and clinical attachment level (adjacent tooth) measured with a standardised UNC-15 probe.
Colorimetric integration | 1 month after surgery, 6 months after surgery
  Colorimetric integration of the augmented buccal peri-implant mucosa, relative to the buccal attached gingiva of the mesial and distal adjacent tooth, quantified throughout the ∆E score, calculated on standardised digital photographs.
Patients related outcome measures | 7 days after surgery, 14 days after surgery, 1 month after surgery, 6 months after surgery
  Patients pain and discomfort with respect to the procedure evaluated with the short form of the McGill pain questionnaire (SF-MPQ).
Microcirculation of the grafted area | before surgery, after surgery, 7 days after surgery, 14 days after surgery, 1 month after surgery, 6 months after surgery
  Microcirculation of the treated area evaluated with a laser Doppler flowmeter.
Morphology of the grafted area | 1 month after surgery or 2 months after surgery or 4 months after surgery or 6 months after surgery
  Descriptive histology performed on paraffin embedded sections from buccal gingival specimens, stained with hematoxylin-eosin.
Revascularization and reinnervation of the grafted area | 1 month after surgery or 2 months after surgery or 4 months after surgery or 6 months after surgery
  Immune histochemistry performed on paraffin embedded, hematoxylin-eosin stained sections using markers of tissue revascularization and reinnervation.
Full mouth Plaque score | baseline, after surgery, 1 month after surgery, 6 months after surgery
  Full muouth plaque score measured with a standardised UNC-15 probe.
Full mouth Bleeding score | baseline, after surgery, 1 month after surgery, 6 months after surgery
  Full mouth bleeding score measured with a standardised UNC-15 probe.
Keratinised tissue width | baseline, after surgery, 1 month after surgery, 6 months after surgery
  Keratinised tissue width measured with a standardised UNC-15 probe.
Bleeding on probing | baseline, after surgery, 1 month after surgery, 6 months after surgery
  Presence/absence of bleeding on probing at the treated implant measured with a standardised UNC-15 probe.
Modified Plaque index | baseline, after surgery, 1 month after surgery, 6 months after surgery
  Presence/absence of plaque at the treated implant

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz Alonso, Study Chair — Faculty of Odontology, University Complutense, Madrid, Spain; David Palombo, Study Director — Faculty of Odontology, University Complutense, Madrid, Spain
Locations (1):
- Department of Periodontology, University Complutense Madrid, Spain, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Result] Chappuis V, Araujo MG, Buser D. Clinical relevance of dimensional bone and soft tissue alterations post-extraction in esthetic sites. Periodontol 2000. 2017 Feb;73(1):73-83. doi: 10.1111/prd.12167. PMID 28000281
- [Result] Johnston WM, Kao EC. Assessment of appearance match by visual observation and clinical colorimetry. J Dent Res. 1989 May;68(5):819-22. doi: 10.1177/00220345890680051301. PMID 2715476
- [Result] McLean TN, Smith BA, Morrison EC, Nasjleti CE, Caffesse RG. Vascular changes following mucoperiosteal flap surgery: a fluorescein angiography study in dogs. J Periodontol. 1995 Mar;66(3):205-10. doi: 10.1902/jop.1995.66.3.205. PMID 7776165
- [Result] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Result] Perotto S, Romano F, Cricenti L, Gotti S, Aimetti M. Vascularization and Innervation of Connective Tissue Grafts in the Treatment of Gingival Recessions: A Histologic and Immunohistochemical Study. Int J Periodontics Restorative Dent. 2017 Jul/Aug;37(4):551-558. doi: 10.11607/prd.3020. PMID 28609502
- [Result] Rojo E, Stroppa G, Sanz-Martin I, Gonzalez-Martin O, Alemany AS, Nart J. Soft tissue volume gain around dental implants using autogenous subepithelial connective tissue grafts harvested from the lateral palate or tuberosity area. A randomized controlled clinical study. J Clin Periodontol. 2018 Apr;45(4):495-503. doi: 10.1111/jcpe.12869. Epub 2018 Feb 23. PMID 29334403
- [Result] Sanz-Martin I, Encalada C, Sanz-Sanchez I, Aracil J, Sanz M. Soft tissue augmentation at immediate implants using a novel xenogeneic collagen matrix in conjunction with immediate provisional restorations: A prospective case series. Clin Implant Dent Relat Res. 2019 Feb;21(1):145-153. doi: 10.1111/cid.12696. Epub 2018 Dec 3. PMID 30508313
- [Result] Tatarakis N, Gkranias N, Darbar U, Donos N. Blood flow changes using a 3D xenogeneic collagen matrix or a subepithelial connective tissue graft for root coverage procedures: a pilot study. Clin Oral Investig. 2018 May;22(4):1697-1705. doi: 10.1007/s00784-017-2261-5. Epub 2017 Oct 27. PMID 29080078
- [Result] Thoma DS, Zeltner M, Hilbe M, Hammerle CH, Husler J, Jung RE. Randomized controlled clinical study evaluating effectiveness and safety of a volume-stable collagen matrix compared to autogenous connective tissue grafts for soft tissue augmentation at implant sites. J Clin Periodontol. 2016 Oct;43(10):874-85. doi: 10.1111/jcpe.12588. Epub 2016 Aug 12. PMID 27310522
- [Result] Thoma DS, Naenni N, Figuero E, Hammerle CHF, Schwarz F, Jung RE, Sanz-Sanchez I. Effects of soft tissue augmentation procedures on peri-implant health or disease: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Mar;29 Suppl 15:32-49. doi: 10.1111/clr.13114. PMID 29498129